CLINICAL TRIAL: NCT02853422
Title: A Study Evaluating The Clinical Utility Of The Health-Related Quality-Of-Life QLQ-GINET21 Questionnaire In The Treatment Of Patients With Gastrointestinal Neuroendocrine Tumours QUALINETS Study
Brief Title: Quality-Of-Life QLQ-GINET21 Questionnaire In The Treatment Of Patients With Gastrointestinal Neuroendocrine Tumours
Acronym: QUALINETS
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-ES-52030-351; IPS-ANT- 2015-01 (Other: Spanish Drug Agency AEMPS)
Record Dates: First submitted 2016-04-28; First posted 2016-08-02 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Gastrointestinal Neuroendocrine Tumours

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the utility of the QLQ-GINET21 in making clinical and therapeutic decisions.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of gastrointestinal endocrine tumour.
* Patient able to read and understand the study questionnaires.
* Patient who has given informed consent in writing to take part in the study.

Exclusion Criteria:

* Patient who is taking part in another clinical study during the study.
* Patients with another serious malignancy.
* Patients unable to meet the requirements of the protocol (non-compliant patients or those unfit to answer the questionnaires).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Survey on the clinical utility of the QLQ-GINET21, which the investigator is to complete for each patient enrolled | Day 1

SECONDARY OUTCOMES:
Socio-demographic variables of the investigator | Day 1
  Descriptive analysis of socio-demographic variables including age, gender, years of experience in treating neuroendocrine tumours (NETs), area of professional activity, capacity of the hospital
Socio-demographic variables of the patient | Day 1
  Descriptive analysis of socio-demographic variables including age, gender, employment status, marital status, educational level
Patients' health-related quality of life concerning gastrointestinal neuroendocrine using QLQ-GINET21 | Day 1
Patients' health-related quality of life concerning gastrointestinal neuroendocrine using QLQ-C30 | Day 1
Clinical characteristics of patients - time since first therapeutic intervention | Day 1
Health status as perceived by the patient | Day 1
  Patients assess their overall health status in relation to their gastrointestinal neuroendocrine tumour, with a question designed for this purpose: "Please answer the question by marking the response that best defines your current health status as related to your neuroendocrine disease". The response options are: Very good, quite good, somewhat good, neither good nor bad, somewhat bad, quite bad, very bad.
Clinical assessment of patient's health status by the investigator | Day 1
  The investigator evaluates the patient's health status in relation to the gastrointestinal neuroendocrine tumour by answering the following question: Overall, how would you rate the patient's health status in relation to their gastrointestinal neuroendocrine tumour as of today? The response options are: Very good, quite good, somewhat good, neither good nor bad, somewhat bad, quite bad, very bad.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (32):
- Portugal (2):
  - Instituto Portuguès de Oncologia de Lisboa, Lisbon
  - Instituto Portuguès de Oncologia do Porto, Porto
- Spain (30):
  - Hospital General Univ. Elche, Alicante
  - Hospital Clinico y Provincial, Barcelona
  - Hospital Univ. Burgos, Burgos
  - Hospital Jerez de la Frontera, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital General Univ. Ciudad Real, Ciudad Real
  - Hospital Univ. de Cabueñes, Gijón
  - ICO Girona, Girona
  - Hospital Can Mises, Ibiza Town
  - Hospital Univ. León, León
  - Hospital de La Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Univ. Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Univ. Puerta del Hierro, Madrid
  - Hospital Regional Univ. Málaga, Málaga
  - Hospital Univ.Virgen de la Victoria, Málaga
  - Hospital Rey Juan Carlos I, Móstoles
  - Hospital General Univ. Morales Meseguer, Murcia
  - Hospital Univ. Son Espases, Palma
  - Hospital Son Llàtzer, Palma
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clínico Univ. Salamanca, Salamanca
  - Hospital Clínico Univ. de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Hospital Univ. Virgen del Rocío, Seville
  - Hospital Univ. Mútua de Terrasa, Terrassa
  - Hospital de Galdakao, Usansolo
  - Hospital Univ. Fe, Valencia
  - Hospital Clínico Univ. Valladolid, Valladolid